CLINICAL TRIAL: NCT05215717
Title: Feasibility of Self-Administered Hypnosis for Sleep Quality for Individuals With Mild Cognitive Impairment
Brief Title: Hypnosis for Sleep Quality for Individuals With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Gary R. Elkins, Director of Mind-Body Medicine Research Lab, Baylor University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 3R01AT009384-05S1 (NIH)
Record Dates: First submitted 2022-01-03; First posted 2022-01-31 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Mild Cognitive Impairment; Poor Quality Sleep
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will be randomized and enrolled into one of two study groups, self-administered hypnosis (treatment group) or sham white noise hypnosis (control group).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Administered Hypnosis (Experimental): Participants randomized to the self-administered hypnosis group will receive five audio-recordings of self-administered hypnosis, specifically targeting sleep improvement, which they will use for daily home practice.
  Interventions: Behavioral: Self-Administered Hypnosis
- White Noise Hypnosis Control (Active Comparator): Participants randomized to the white noise hypnosis control will receive the same information and contact with the therapist but will be provided with audio recordings that contain white noise as a sham hypnosis condition. These recordings include instructions and the use of white noise as a hypnotic induction.
  Interventions: Behavioral: Self-Administered White Noise Hypnosis

INTERVENTIONS:
Behavioral: Self-Administered Hypnosis — Participants randomized to the self-administered hypnosis group will receive five audio-recordings of self-administered hypnosis, specifically targeting sleep improvement, which they will use for daily home practice.
  Arms: Self-Administered Hypnosis
Behavioral: Self-Administered White Noise Hypnosis — Participants randomized to the white noise hypnosis control will receive the same information and contact with the therapist, but will be provided with audio recordings that contain white noise as a sham hypnosis condition. These recordings include instructions and the use of white noise as a hypnotic induction.
  Arms: White Noise Hypnosis Control

SUMMARY:
With the long-range goal to identify an efficacious and practical intervention to improve sleep for individuals with MCI, this pilot study will enroll 20 individuals with MCI into either a self-administered hypnosis for sleep program or a sham white noise hypnosis program. Participants will practice hypnosis delivered via audio recording once per day in their own home for 7 weeks. Upon completion of the study, insight will be gained regarding accrual, retention, and feasibility of the intervention and measures. Data from this pilot study is essential to inform and plan a future R01 proposal to determine the efficacy of the self-administered hypnosis intervention to improve sleep quality and duration, as well as other benefits, with individuals with mild cognitive impairment.

DETAILED DESCRIPTION:
Study Objectives

Aim 1: Determine the accrual, retention, adherence and feasibility, and randomization to the self-administered hypnosis program among individuals with MCI. Feasibility will be determined by (1) drop-out rate, (2) participants' rating of the program, and (3) participants' rating of treatment satisfaction. Adherence will be determined through at-home practice logs. Essential experience on accrual and retention data as well.

Aim 2: Determine feasibility of measures: PSQI, actigraphy recordings, and sleep diaries to assess sleep quality and duration, as well as feasibility of secondary self-report outcome measures of insomnia severity, stress, cognition, and pain among individuals with MCI.

Aim 3: Determine perceptions of hypnosis and potential barriers for the MCI population and feedback.

Participant Selection and Recruitment Plan

A sample of approximately 20 individuals with mild cognitive impairment, both male and female, who suffer from poor sleep will be enrolled in the study. A screening checklist will be used for screening participants who are interested.

Potential participants will be identified (1) via advertisements and press releases, (2) via physician and health care provider referral, support groups (3) and (4) targeted mailings. Participant's eligibility will be determined by criteria listed on a screening checklist. The investigator has used these strategies in prior studies and has demonstrated ability to accrue the required number of participants.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of MCI (a score of less than or equal to 3 on the Memory Complaint Scale30) and a score between 7-18 on the Montreal Cognitive Assessment (MoCA) - BLIND Version 8.121
* Self-reported sleep duration of less than or equal to 6 hours per day/night as indicated on the PSQI
* Signed informed consent

Exclusion Criteria:

* Use of any prescription or over-the-counter therapy for sleep
* Severe or unstable medical or psychiatric illness
* Current use of hypnosis for any condition
* Inability to speak or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2022-11-06 (Actual)

PRIMARY OUTCOMES:
Daily At-home Self-Hypnosis Practice Log | Through study completion, an average of 7 weeks
  All participants will be given guidance on the use of hypnosis and recordings for at-home practice throughout the study. Participants will be instructed in daily practice of hypnosis and asked to keep a daily at-home self-hypnosis practice form during the intervention period. Adherence will be assessed via calculation of participants' frequency of hypnosis practice from these daily hypnosis practice forms. The participant will be asked to practice daily and to complete a practice log, recording the frequency of practice of self-administered hypnosis. Practice logs will be used to assess frequency of practice.
Program Rating Scale | One week
  In order to assess participants' perceptions of the value of the hypnosis program they receive, they will be asked "How do you rate this hypnosis program overall in regard to ease of use?" and "How do you rate this hypnosis program overall in regard to improving your sleep?" Responses will be given on a 10-point scale ranging from 1 (Poor) to 10 (Excellent) at follow-up.
Treatment Satisfaction Scale | One week
  Participants will be asked to rate their overall level of satisfaction with the intervention. A 10-point VAS scale anchored with 0 "Completely Dissatisfied" to 10 "Completely Satisfied" will be given at follow-up.
Wrist Actigraphy - Objective Sleep Duration | Up to 2 weeks
  Wrist actigraphy is a widely used and well-validated measure of sleep duration. Participants will be asked to wear an actigraph (Actiwatch 2; Phillips Respironics, Andover, MA), resembling a wristwatch, on their non-dominant wrist. A motion detection device located within the actigraph records movement. After data is collected and stored within the actigraph it can be analyzed with the Philips Respironics 5 software program.
  This program uses a series of logarithms to measure various factors associated with sleep quality, such as total sleep duration, sleep efficiency, sleep onset latency, and the number of times participants woke during the night. Each of these factors will be combined to assess and report objective sleep duration in hours per day/night for participants. For the present study, participants will be asked to wear the actigraph for one week at baseline and for one week at follow-up.
Pittsburgh Sleep Quality Index | Up to 2 weeks
  Participants will be asked to complete the Pittsburgh Sleep Quality Index (PSQI) during screening and at follow-up. The PSQI is a 19-item self-report inventory designed to measure sleep quality. The 19 items are grouped into 7 subscales: 1) sleep quality, 2) sleep efficiency, 3) daytime dysfunction, 4) sleep latency, 5) sleep disturbances, 6) sleep duration, and 7) use of sleep medication. These seven subscales are scored on a scale of 0-3 with higher scores indicating greater sleep pathology. Cronbach's alphas for the PSQI range from .70 to .80.
Daily Sleep Diaries | Through study completion, an average of 7 weeks
  A daily sleep diary where participants record time awake and time to bed will be used. Participants will be asked to complete a daily sleep diary upon awakening each morning for a week at baseline, daily during the intervention weeks, and a week at follow-up.
Epworth Sleepiness Scale | Through study completion, an average of 7 weeks
  Participants will be asked to complete the Epworth Sleepiness Scale (ESS) during baseline and at follow-up. The ESS is an 8-item self-report measure that asks participants to indicate how likely they are to fall asleep while engaging in eight different everyday activities (e.g., watching television, sitting in traffic). Items are scored on a scale from 0-3 with higher scores indicating a greater probability of falling asleep. Previous research indicates that the ESS has a Cronbach's alpha of .88
Sleep Environment Questionnaire | Through study completion, an average of 7 weeks
  Participants will be asked to complete the Sleep Environment Questionnaire during baseline and at follow-up. The Sleep Environment Questionnaire is an 11- item self-report measure that asks about the environment in which a person sleeps. Response options include "True," "False," or "Not Applicable."
Attitudes Toward Hypnosis Scale | Through study completion, an average of 7 weeks
  The 14-item Attitudes Toward Hypnosis Scale will be used to assess attitudes toward hypnosis at baseline and at follow-up. This scale has shown internal consistency in previous studies, Cronbach's alpha = .81. A total attitude toward hypnosis score will be calculated for each participant by summing scores across the 14 items with higher scores indicating more positive attitudes toward hypnosis.

SECONDARY OUTCOMES:
Insomnia Severity Index | Through study completion, an average of 7 weeks
  Participants will be asked to complete the Insomnia Severity Index (ISS) at baseline and follow-up. The ISI consists of seven items that measure the severity of sleep onset, sleep maintenance, and early morning awakening problems, as well as the participant's satisfaction with her current sleep pattern, the extent to which lack of sleep interferes with daily functioning, how noticeable this impairment is to other people, and the extent to which the participant is worried or distressed about their lack of sleep. Items are scored on a scale from 0-4 with total score of 15 or higher indicating the presence of clinical insomnia24. Past research indicates that internal reliability estimates for the ISI range from .74 to .78.
Perceived Stress Scale | Through study completion, an average of 7 weeks
  The Perceived Stress Scale (PSS) will be used to measure stress at baseline and follow-up. The PSS includes 14 items that assess levels of perceived stress and to what degree individuals perceive events in their life as stressful during the previous month. Higher scores indicate greater stress. Past research indicates that Cronbach's alpha for the PSS is .85.
PROMIS Cognitive Function - Short Form | Through study completion, an average of 7 weeks
  Cognition will be assessed at baseline and at follow-up using the PROMIS Cognitive Function - Short Form Scale. This scale includes 8 items and measures self-reported cognitive functioning during the past 7 days. Items are scored from a scale of 1 (Very Often) to 5 (Never). Items are summed to create a total score and higher scores indicate better cognitive functioning.
Pain Visual Analog Scale | Through study completion, an average of 7 weeks
  Participants will be asked to rate their pain on a 100-mm visual analog scale (VAS) during baseline and follow-up. Participants will be asked to place an "x" along the 100-mm line to indicate the severity of their pain over the past week, with the lower end of the scale being anchored by the phrase "no pain" and the upper end of the scale being anchored by the phrase "the most intense pain possible."
Motivation Scale | One week during baseline week
  Motivation to use hypnosis is an important factor to be assessed. Motivation to use hypnosis to improve sleep quality will be assessed at baseline using a numerical rating scale that states, "How motivated are you to use hypnosis to improve sleep?" This item will be rated on a scale of 1 (Not Motivated at All) to 10 (Very Motivated).

OTHER OUTCOMES:
Post-Participation Interview | 1 week
  In order to gather qualitative data to improve future studies, participants will be asked to participate in a post-participation interview. An experienced and trained doctoral student will conduct interviews and create summary statements regarding topics including ease of use of the intervention, barriers of using the audio recordings, finding the time to practice, and improvement of the intervention. Interviews will be recorded, and transcripts will be typed out.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor University, Waco, Texas, United States